CLINICAL TRIAL: NCT03224455
Title: Environmental Risk Factors for Pediatric Sleep Disordered Breathing
Brief Title: Environmental Assessment of Sleep in Youth
Acronym: EASY
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Wanda Phipatanakul, Professor of Pediatrics, Harvard Medical School (HMS and HSDM)
Other Study IDs: IRB-P00025433
Record Dates: First submitted 2017-07-17; First posted 2017-07-21 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Sleep Disorders in Children; Environmental Exposure
Keywords: sleep; sleep in children; children and sleep; environment; environment and sleep; environment and children

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this research study, investigators want to learn more about the factors that influence children's breathing during sleep and their sleep quality. Specifically, investigators are interested in factors that are related to risk of snoring, sleep apnea (a condition where breathing stops during sleep), and poor sleep quality.

DETAILED DESCRIPTION:
Investigators are doing a research study to gather information to help better understand why snoring and sleep problems are so common in the community, and how the home and neighborhood environment impacts sleep in children. Investigators want to know if factors such as the quality of air, household dust, environmental noise, and family routines impact sleep and other health and behavioral factors associated with sleep.

Investigators want to test how sleep is influenced by factors such as: the quality of air inside and outside the child's home (including measuring pollution, second hand smoke, and dust); temperature and humidity; family routines and interactions; and characteristics of the home. Investigators will ask participants to come in for a one time visit for undergoing procedures as well as answering questions regarding general health, asthma and sleep. 10% of the participating children will have a second home assessment and sleep monitoring procedures performed 6 months after the initial home assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age 6-12 years
* Children living (50% of the time or more) at their current residence for at least 1 month

Exclusion Criteria:

* Children with severe chronic diseases (e.g. cancer, genetic or congenital disorders interfering with mobility)
* Children with severe neurobehavioral, neurodevelopmental or psychiatric disorders requiring special assistance
* Children living in the current residence for < 1 month will be not be eligible.
* Families who do not speak English or Spanish well enough to complete the neuropsychological measures, as validated versions in other languages are not available for all of the measures.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children 6-12 years old who live in the Boston area.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-17 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index (AHI) | 2 days
  Oxygen Desaturation Index (ODI; >3%desaturation dips) registered in the WatchPAT. Estimated Apnea and Hypopnea Indices, % recording time snoring using the EMFIT QS under mattress sensor.
Apnea Hypopnea Index (AHI) | 7days
  Estimated Apnea and Hypopnea Indices, % recording time snoring using the EMFIT QS under mattress sensor.

SECONDARY OUTCOMES:
sleep duration and sleep efficiency | 7 days
  average of the sleep sensor readings
Sleepiness Quality of Life | 7 days
  total score of Epworth Sleepiness Scale(ESS)
Quality of Life score | 7 days
  total score of Pediatric Quality of Life (PedsQL) (0-100) 100 is better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Wanda Phipatanakul, MS. MS., Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No